CLINICAL TRIAL: NCT06315920
Title: Parecoxib Versus Morphine in Acute Pain Management for Sickle Cell Disease Patients in Emergency Department: a Randomized Controlled Trial.
Brief Title: Analgesic Effect of Parecoxib Versus Morphine in SCD Patients Presenting to the Emergency Department
Acronym: PASC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Collaborators: Armed Forces Hospital, Oman (Unknown)
Responsible Party: Principal Investigator, Usama Al-Khalasi, EM Specialist, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFMS-MREC 009/2021
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Sickle-Cell Disease with Crisis
Keywords: SCD, Parecoxib , Opioids
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — parecoxib; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking process involves the following steps:
  Preparation of Medication: A nurse, who is not involved in the direct care or assessment of the patients, will prepare the medications. This nurse is the only individual aware of the specific treatment being administered to each patient. The medications are prepared in a manner that makes them indistinguishable from each other in appearance, labeling, and administration method.
  Administration of Medication: The medications are then administered to the patients by healthcare providers who are blinded to the nature of the medication. This ensures that their assessment of the patient's response is not influenced by knowledge of the treatment being given.
  Assessment and Data Collection: The assessment of pain relief, side effects, and other relevant clinical outcomes is conducted by healthcare providers who are blinded to the treatment allocation. This minimizes bias in the evaluation of the treatment's efficacy and safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parecoxib (Experimental): 40mg of IV Parecoxib
  Interventions: Drug: Parecoxib
- Morphine (Active Comparator): 5 mg of IV Morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Parecoxib — Single dose of 40mg of IV Parecoxib.
  Other Names: a COX-2 selective nonsteroidal anti-inflammatory drug (NSAID)
  Arms: Parecoxib
Drug: Morphine — Single dose of 5 mg of IV Morphine.
  Other Names: Morphine Sulfate
  Arms: Morphine

SUMMARY:
Introduction: This study focuses on the treatment of painful crises in Sickle Cell Disease (SCD) patients using Paracoxib, a non-opioid, compared to Morphine. It addresses the need for alternative medications that reduce opioid dependency while providing effective analgesia.

Objectives:

Primary: Evaluate the analgesic effect of Paracoxib versus Morphine in SCD vaso-occlusive crises.

Secondary: Reduce opioid use/dependence, decrease the length of hospital stays, and monitor side effects related to Paracoxib.

Methodology: A double-blinded randomized controlled trial, conducted in a tertiary care emergency department. The study includes adult SCD patients with moderate to severe crises, excluding non-VOC pain, certain medications, and specific medical conditions. The sample size is 226 patients, split equally into two groups.

Intervention: Patients receive either Morphine or Paracoxib, with periodic assessment of vital signs and pain. Additional Morphine is administered if required. Data collection and analysis are meticulously planned.

Expected Outcomes: Improvement in SCD pain management, reduction in opioid usage, and potential benefits in terms of hospital stays and patient satisfaction.

DETAILED DESCRIPTION:
Introduction: Sickle Cell Disease (SCD) is a prevalent hematological disorder in Oman. Patients frequently present to Emergency Departments (ED) with painful crises, often requiring high doses of opioids like Morphine. However, the complications associated with opioid use, including dependency, necessitate exploring alternative analgesic options. This research proposes a comparative study of Parecoxib, a non-steroidal anti-inflammatory drug (NSAID), and Morphine in managing pain for SCD patients in the ED.

Background: Recent studies have highlighted Parecoxib's potential in various clinical settings. In trauma patients, Parecoxib demonstrated comparable analgesic efficacy to Morphine, suggesting its broader applicability in the ED. Parecoxib has shown benefits in post-operative pain management, reducing opioid requirements and associated adverse events. Notably, in post knee replacement surgeries, Parecoxib effectively managed pain and facilitated functional recovery. It also contributed to decreased postoperative delirium in elderly patients undergoing hip or knee replacement surgery without increasing adverse events.

Research Objectives: The primary objective of this study is to evaluate the analgesic efficacy of Parecoxib versus Morphine in SCD patients experiencing vaso-occlusive crises. Secondary objectives include assessing the potential reduction in opioid dependence, length of hospital stay, recurrence of ED visits, and monitoring any Parecoxib-related side effects in SCD patients.

Methodology:

* Study Design: A double-blinded, randomized controlled trial.
* Study Setting: AFH Emergency Department, a tertiary care institution.
* Target Population: Adult SCD patients (>18 years) presenting with moderate to severe vaso-occlusive crises.
* Exclusion Criteria: Include non-VOC pain, weight < 50 kg, frequent ED visits, recent opioid/NSAID use, contraindications to NSAIDs, lactating mothers, and recent visits to other health institutions.
* Sample Size: The sample size of 226 patients, split into two groups of 113 each, was determined for a two-sided hypothesis test with a 5% significance level and 90% power. This design ensures a high probability of detecting a significant difference in the analgesic efficacy between Parecoxib and Morphine for SCD patients. The calculated size is based on expected effect sizes from previous research, with additional allowance for potential dropouts, ensuring the study's statistical validity and comprehensiveness.
* Intervention: Computer-randomized administration of Morphine or Parecoxib. Continuous monitoring of vital signs and pain assessment at set intervals post-medication administration. Senior emergency physicians and residents will conduct assessments.
* Data Collection and Analysis: The study will be double-blinded, with only the preparing nurse aware of the medication used. Data will be recorded using Epi-Data and analyzed using SPSS version 25.

Expected Outcomes: The study aims to enhance pain management protocols for SCD patients in the ED. By introducing Parecoxib as an alternative to opioids, we anticipate reduced opioid use, shortened hospital stays, fewer ED visits, and overall cost-effectiveness in managing SCD pain crises. The findings will be disseminated through local and international conferences and journals.

ELIGIBILITY:
Inclusion Criteria:

* An adult (>18 years) sickle cell disease patient presents with moderate-severe vaso-occlusive crisis (VOC) to the ED.

Exclusion Criteria:

* Non-VOC Pain (e.g. Acute chest syndrome, sequestration, septic arthritis, Etc.)
* Weight less than 50 KG
* Recurrent visits > one visit/ week
* Opioids within 24hrs
* NSAIDs within 24hrs
* Contraindications to NSAIDs (e.g. allergy, Asthma, CKD, pregnancy, Etc.)
* Lactating mothers
* Visited another health institution within 24hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction at 60 mins. | 60 mintues
  analgesics effect of Parecoxib versus Morphine in sickle cell disease vaso- occlusive crisis.

SECONDARY OUTCOMES:
Adverse Events/Side Effects | 48 hours
  Any reported adverse events reported by subjects or attending doctor
The need of rescue pain medications | 60 mintues
  After 60 min , patients can have rescue medications as standard of care.
Recurrent visit | 48 hours
  Any recurrent visit with painful vaso- occlusive crisis

CONTACTS AND LOCATIONS:
Overall Officials: USAMA ALKHALASI, MD, Study Chair — Armed Forces Hospital, Oman; Muzna Al Sawafi, MD, Principal Investigator — Armed Forces Hospital, Oman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baharuddin KA, Rahman NH, Wahab SF, Halim NA, Ahmad R. Intravenous parecoxib sodium as an analgesic alternative to morphine in acute trauma pain in the emergency department. Int J Emerg Med. 2014 Jan 3;7(1):2. doi: 10.1186/1865-1380-7-2. PMID 24386899
- [Background] Laoruengthana A, Rattanaprichavej P, Reosanguanwong K, Chinwatanawongwan B, Chompoonutprapa P, Pongpirul K. A randomized controlled trial comparing the efficacies of ketorolac and parecoxib for early pain management after total knee arthroplasty. Knee. 2020 Dec;27(6):1708-1714. doi: 10.1016/j.knee.2020.10.005. Epub 2020 Nov 13. PMID 33197808
- [Background] Stoltz RR, Harris SI, Kuss ME, LeComte D, Talwalker S, Dhadda S, Hubbard RC. Upper GI mucosal effects of parecoxib sodium in healthy elderly subjects. Am J Gastroenterol. 2002 Jan;97(1):65-71. doi: 10.1111/j.1572-0241.2002.05265.x. PMID 11808971
- [Background] Rasmussen GL, Steckner K, Hogue C, Torri S, Hubbard RC. Intravenous parecoxib sodium foracute pain after orthopedic knee surgery. Am J Orthop (Belle Mead NJ). 2002 Jun;31(6):336-43. PMID 12083587
- [Background] Zhuang Q, Tao L, Lin J, Jin J, Qian W, Bian Y, Li Y, Dong Y, Peng H, Li Y, Fan Y, Wang W, Feng B, Gao N, Sun T, Lin J, Zhang M, Yan S, Shen B, Pei F, Weng X. Postoperative intravenous parecoxib sodium followed by oral celecoxib post total knee arthroplasty in osteoarthritis patients (PIPFORCE): a multicentre, double-blind, randomised, placebo-controlled trial. BMJ Open. 2020 Jan 9;10(1):e030501. doi: 10.1136/bmjopen-2019-030501. PMID 31924632
- [Background] Mu DL, Zhang DZ, Wang DX, Wang G, Li CJ, Meng ZT, Li YW, Liu C, Li XY. Parecoxib Supplementation to Morphine Analgesia Decreases Incidence of Delirium in Elderly Patients After Hip or Knee Replacement Surgery: A Randomized Controlled Trial. Anesth Analg. 2017 Jun;124(6):1992-2000. doi: 10.1213/ANE.0000000000002095. PMID 28525512
- [Background] Nong L, Sun Y, Tian Y, Li H, Li H. Effects of parecoxib on morphine analgesia after gynecology tumor operation: a randomized trial of parecoxib used in postsurgical pain management. J Surg Res. 2013 Aug;183(2):821-6. doi: 10.1016/j.jss.2013.02.059. Epub 2013 Mar 30. PMID 23587455